CLINICAL TRIAL: NCT05939791
Title: The Effect of Physical Exercise and Dairy Probiotics (Lactobacillus Casei) on Gut Microbiome in Childhood Cancer Survivors
Brief Title: Physical Exercise and Dairy Probiotics in Childhood Cancer Survivors
Acronym: Exerbioall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-0047
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
Keywords: Physical Exercise, Gut Microbiome, Exercise Training, Veillonella
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): Children previously diagnosed and treated for acute lymphoblastic leukemia in remission between 1 and 3 years with physical exercise intervention
  Interventions: Other: Lacticaseibacillus paracasei subsp. Paracasei CNCMI-1518; Other: Physical exercise
- Passive (No Intervention): Children previously diagnosed and treated for acute lymphoblastic leukemia in remission between 1 and 3 years without physical exercise intervention

INTERVENTIONS:
Other: Lacticaseibacillus paracasei subsp. Paracasei CNCMI-1518 — The commercial probiotic dairy product has been provided to PALL along with physical training once a day for 8 weeks. Each serving contained 20 billion CFUs of Lacticaseibacillus paracasei subsp. Paracasei CNCMI-1518 (Lactobacillus casei CNCMI-1518). Each patient's legal representative was advised to follow a normal diet when preparing and providing food for children.
  Arms: Exercise training
Other: Physical exercise — The individual online (MS Teams) training program for PALL in the length of 8 weeks included 25-45 minutes of moderate-to-vigorous physical exercise, twice a week, under the supervision. The structure of the exercise program was developed to improve endurance and gradually rebuild muscular strength. The exercise program's structure was created to increase endurance and gradually rebuild muscular strength. Large muscle groups were the focus of training sessions, which also placed a strong emphasis on proper technique. A strength exercise squat was given consideration as a movement required to meet necessities. (e.g., sitting or standing). Each exercise consisted of between 10 and 15 repetitions in each series and 2 to 3 series overall.
  Arms: Exercise training

SUMMARY:
The goal of this clinical trial is to to compare the structure of the intestinal microbiome between children shortly after treatment for acute lymphoblastic leukemia (1-3 years after cancer treatment) and healthy controls. And then to provoke a positive shift of bacterial diversity by physical activity and probiotics in cured pediatric oncology patients with persistent gut microbiome disruptions.

The main question[s] it aims to answer are:

* Are differences in bacterial richness between healthy controls and pediatric oncology patients ≥12 months after cancer treatment apparent?
* Has the combination of physical exercise and probiotics had a positive influence on the structure of the gut microbiome in childhood cancer survivors in remission? Two times per week of physical activity and daily dairy consumption with probiotics will be required of participants for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

- children previously diagnosed and treated for acute lymphoblastic leukemia in remission between 1 and 3 years

Exclusion Criteria:

* acute respiratory infection during intervention
* more than 20% skipped exercise training sessions

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The shift of gut microbiome by physical exercise and consumption of dairy probiotics. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Hematology National Institute of Children's Diseases Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No